CLINICAL TRIAL: NCT03473652
Title: Feasibility of Adapted Physical Activity Based on a Walking Platform in Hospitalized Old Patients for Cancer
Acronym: APPAHOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APPAHOCA
Record Dates: First submitted 2018-03-12; First posted 2018-03-22 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Oncology; Adapted Physical Activity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted walking platform (Other)
  Interventions: Other: Adapted walking platform

INTERVENTIONS:
Other: Adapted walking platform — The walking sessions will be carried out on a suitable walking platform, including a connected play tablet.

SUMMARY:
The investigator propose to evaluate the interest of the provision of a suitable treadmill offering fall protection and verticalization assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer
* Patient over 70 years old hospitalized 48 hours or more
* Patient identified as eligible for medical prescription of Adapted physical activity
* Mastery of the French language ;
* Patient affiliated to a social security scheme
* Patient giving written consent

Exclusion Criteria:

* Patient totally unable to communicate
* Patient in terminal palliative care
* Patient with a size <1m35 or> 2m and / or a weight> 130kg
* Patient unable to perform Adapted physical activity sessions
* Patient unable to wear a restraint harness.
* Patient deprived of liberty or under guardianship
* Patient unable to comply with protocol requirements for geographical, social or psychopathological reasons

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - CHU, Caen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adapted walking platform: After a daily medical assessment of the walking capacities, patients were invited to use the Ema walking platform for 6 to 30 minutes. A health physical activity teacher brought the patients to the walking platform using a whellchair. He installed and assisted the patient during the training session while maintaining the required hygienic conditions.
Period: Overall Study
Arm/Group | Adapted walking platform
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 45 patients were included.
Arm/Group | Adapted Walking Platform
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Living place [Count of Participants; unit: Participants] — Patients were asked if they were living in a nursing home, a senior residence of individual home.
  Participants
    Nursing home | 1
    Senior residence | 1
    Individual home | 43

OUTCOME MEASURES:

1. Primary Outcome: Patient Adherence to Use a Walking Platform
Description: Adapted physical activity on a walking platform will be considered feasible if > or = to 70% of patients perform > or = to 2 sessions of 6 minutes or more during hospitalization for cancer lasting > or = to 48h
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Adapted walking platform
Number analyzed (Participants) | 45
Participants | 26

ADVERSE EVENTS:
Time Frame: Not collected
Description: Not collected
Arm/Group | Adapted walking platform
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT03473652/Prot_000.pdf